CLINICAL TRIAL: NCT01056315
Title: A Randomized, Multicenter, Double-blind, Placebo-controlled, Parallel-group Trial to Assess the Analgesic Efficacy and Safety of a New Analgesic Compared to Placebo in Subjects With Painful Diabetic Peripheral Neuropathy
Brief Title: A Trial in Painful Diabetic Peripheral Neuropathy With GRT3983Y
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was stopped due to difficult enrolment
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 131885
Record Dates: First submitted 2009-12-21; First posted 2010-01-26 (Estimated); Results first posted 2012-05-03 (Estimated); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Analgesia; Diabetic Neuropathy; Neuropathic pain; Painful; Chronic pain
MeSH Terms: conditions — Diabetic Neuropathies; Agnosia; Neuralgia; Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A GRT3983Y (Experimental): Participants randomly assigned to receive GRT3983Y.
  Interventions: Drug: GRT3938Y
- B Placebo (Placebo Comparator): Participants randomly assigned to placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GRT3938Y — Overencapsulated tablets of GRT3983Y, 100 to 300mg daily dose, 16 weeks treatment.
  Arms: A GRT3983Y
Drug: Placebo — Overencapsulated tablets of placebo, 16 weeks treatment.
  Arms: B Placebo

SUMMARY:
This trial is assessing the analgesic efficacy and safety of a new central analgesic in subjects with pain due to diabetic peripheral neuropathy (DPN).

ELIGIBILITY:
Inclusion Criteria:

* Symmetrical painful diabetic peripheral neuropathy

Exclusion Criteria:

* History of hypersensitivity, allergy or contraindication to opioids and acetaminophen
* Confounding painful conditions
* Significant vascular disease
* History or risk of seizure
* Chronic disease that might effect drug absorption, distribution, metabolism, or excretion
* Female subjects who are being pregnant or breastfeeding
* Evidence or history of alcohol, medication, or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Grünenthal GmbH
Locations (61):
- United States (61):
  - Site 127, Fairhope, Alabama
  - Site 130, Homewood, Alabama
  - Site 112, Tucson, Arizona
  - Site 129, Escondido, California
  - Site 209, Fullerton, California
  - Site 135, Long Beach, California
  - Site 202, Northridge, California
  - Site 208, Northridge, California
  - Site 219, Northridge, California
  - Site 203, San Francisco, California
  - Site 116, Santa Ana, California
  - Site 118, Santa Ana, California
  - Site 121, Santa Ana, California
  - Site 133, Santa Ana, California
  - Site 126, Vista, California
  - Site 214, Vista, California
  - Site 201, Waterbury, Connecticut
  - Site 136, Deerfield Beach, Florida
  - Site 137, Deerfield Beach, Florida
  - Site 140, Deerfield Beach, Florida
  - Site 216, Deerfield Beach, Florida
  - Site 217, Deerfield Beach, Florida
  - Site 218, Deerfield Beach, Florida
  - Site 117, Fort Myers, Florida
  - Site 124, Jacksonville, Florida
  - Site 228, Jupiter, Florida
  - Site 101, Orlando, Florida
  - Site 226, Orlando, Florida
  - Site 206, Sarasota, Florida
  - Site 212, West Palm Beach, Florida
  - Site 142, Atlanta, Georgia
  - Site 128, Chicago, Illinois
  - Site 223, Chicago, Illinois
  - Site 114, Leawood, Kansas
  - Site 102, Paducah, Kentucky
  - Site 211, Baltimore, Maryland
  - Site 108, East Bridgewater, Massachusetts
  - Site 113, Las Vegas, Nevada
  - Site 122, Princeton, New Jersey
  - Site 230, New York, New York
  - Site 109, Rochester, New York
  - Site 225, Asheville, North Carolina
  - Site 115, High Point, North Carolina
  - Site 227, Canton, Ohio
  - Site 233, Cincinnati, Ohio
  - Site 111, Toledo, Ohio
  - Site 125, Toledo, Ohio
  - Site 104, Philadelphia, Pennsylvania
  - Site 106, Philadelphia, Pennsylvania
  - Site 205, Philadelphia, Pennsylvania
  - Site 105, Austin, Texas
  - Site 213, Corpus Christi, Texas
  - Site 110, Houston, Texas
  - Site 123, Houston, Texas
  - Site 204, Houston, Texas
  - Site 210, Houston, Texas
  - Site 231, Houston, Texas
  - Site 131, San Antonio, Texas
  - Site 215, San Antonio, Texas
  - Site 221, San Antonio, Texas
  - Site 139, Provo, Utah

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 503 participants were excluded from the trial before assignment to a treatment group because they did not meet the inclusion and or exclusion criteria.
Period: Overall Study
Arm/Group | GRT3983Y | Placebo
Started | 27 | 23
Completed | 13 | 12
Not Completed | 14 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GRT3983Y | Placebo | Total
Number analyzed (Participants) | 27 | 23 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 14 | 34
  >=65 years | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.38 (8.942) | 60.27 (10.438) | 59.79 (9.568)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  United States | 27 | 23 | 50

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Intensity
Description: The primary efficacy endpoint is the change from baseline in the mean of the daily average pain intensity scores (on an 11-point NRS) over the last 7 days of the 12-week maintenance (Week 16).
Time Frame: Baseline; last 7 days of 12-week maintenance
Population: Efficacy data were not analyzed because of the limited number of subjects with efficacy data at the time of the early termination of the trial.
Groups:
- GRT3983Y: Participants randomly assigned to receive GRT3983Y.
- Placebo: Participants randomly assigned to receive placebo.
Arm/Group | GRT3983Y | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in the Mean of the Daily Average Pain Intensity Scores (on an 11-point NRS) Over the Entire 12-week Maintenance
Time Frame: Baseline, Daily scores over entire 12 week maintenance
Population: as for outcome 1
Arm/Group | GRT3983Y | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Proportion of Subjects Achieving Various Levels of Pain Improvement (Including 30% and 50%) Based on the Percent Change From Baseline to the Last 7 Days of the 12-week Maintenance on an 11-point NRS (Responder Analysis).
Time Frame: Baseline, Last 7 days of 12-week maintenance
Population: as for outcome 1
Arm/Group | GRT3983Y | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in the Mean of the Daily Average Pain Intensity Scores (on an 11-point NRS) Over Each Week of Maintenance.
Time Frame: Baseline; daily scores over each week of maintenance
Population: as for outcome 1
Arm/Group | GRT3983Y | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline of the Weekly Mean of Night Pain Intensity (on an 11-point NRS).
Time Frame: Baseline; weekly mean
Population: as for outcome 1
Arm/Group | GRT3983Y | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline of the Weekly Mean of Current Pain Intensity (on an 11-point NRS) in the Evening and in the Morning, Respectively.
Time Frame: Baseline, weekly mean
Population: as for outcome 1
Arm/Group | GRT3983Y | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Brief Pain Inventory Scores: Changes From Baseline to Day 8, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71, Day 85, Day 99, and Day 113 (Final Visit).
Time Frame: Baseline, weekly mean
Population: as for outcome 1
Arm/Group | GRT3983Y | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Neuropathic Pain Symptoms Inventory: Changes From Baseline to Day 8, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71, Day 85, Day 99 and Day 113 (Final Visit)
Time Frame: Baseline, weekly mean
Population: as for outcome 1
Arm/Group | GRT3983Y | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Patient Global Impression of Change Using a 7-point Verbal Rating Scale, on Day 29, Day 71 and Day 113 (Final Visit).
Time Frame: Day 29, Day 71 and Day 113.
Population: as for outcome 1
Arm/Group | GRT3983Y | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Short Form 36 Health Survey (SF-36®): Changes From Baseline to Day 29, Day 71 and Day 113 (Final Visit).
Time Frame: Baseline, Day 29, Day 71 and Day 113.
Population: as for outcome 1
Arm/Group | GRT3983Y | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: EuroQol-5 Dimension Health Questionnaire: Changes From Baseline to Day 29, Day 71 and Day 113 (Final Visit).
Time Frame: Baseline, Day 29, Day 71 and Day 113.
Population: as for outcome 1
Arm/Group | GRT3983Y | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Assessment of Each Item of the Leeds Sleep Evaluation Questionnaire: Changes From Baseline to Day 29, Day 71 and Day 113 (Final Visit).
Time Frame: Baseline, Day 29, Day 71 and Day 113.
Population: as for outcome 1
Arm/Group | GRT3983Y | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Hospital Anxiety and Depression Scale: Changes From Baseline to Day 29, Day 71 and Day 113 (Final Visit).
Time Frame: Baseline, Day 29, Day 71 and Day 113.
Population: as for outcome 1
Arm/Group | GRT3983Y | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Time to Treatment Discontinuation Due to Lack of Efficacy.
Time Frame: Baseline to time to treatment discontinuation
Population: as for outcome 1
Arm/Group | GRT3983Y | Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Assessment of Rescue Medication Usage During the 4-week Titration.
Time Frame: 4-week titration phase
Population: as for outcome 1
Arm/Group | GRT3983Y | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | GRT3983Y | Placebo
Serious Adverse Events (participants affected / at risk) | 2/27 | 1/23
Other Adverse Events (participants affected / at risk) | 15/27 | 14/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GRT3983Y (N=27) | Placebo (N=23)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GRT3983Y (N=27) | Placebo (N=23)
Nausea (Gastrointestinal disorders) | 10 (13) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1)
Somnolence (Nervous system disorders) | 4 (5) | 1 (2)
Headache (Nervous system disorders) | 3 (4) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
No participants were analyzed as the study was terminated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is the Institution and Principal Investigator's obligation not to publish any information declaration, invention or whatsoever which is in connection with this Agreement without the prior written consent of the Sponsor.